CLINICAL TRIAL: NCT00278590
Title: Allogeneic Stem Cell Transplantation in Patients With Systemic Lupus Erythematosus
Brief Title: Allogeneic Stem Cell Transplantation in Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DI SLE.Allo2004
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- allogeneic stem cell transplantation (Experimental): allogeneic stem cell transplantation will be performed
  Interventions: Biological: Allogeneic Stem Cell Transplantation

INTERVENTIONS:
Biological: Allogeneic Stem Cell Transplantation — Allogeneic stem cell transplantation will be performed.

SUMMARY:
This trial is designed to evaluate the safety of treating systemic lupus erythematosus participants with cyclophosphamide and CAMPATH-1H followed by allogeneic stem cell transplant. There will be no randomization in this study. All subjects who are determined to be eligible for the study treatment will receive cyclophosphamide and CAMPATH-1H followed by allogeneic stem cell transplant. The purpose of the intense chemotherapy is to destroy the cells in the immune system which may be causing this disease. The purpose of the stem cell infusion is to produce a normal immune system that will no longer attack body. The study purpose is to examine whether this treatment will result in improvement in the lupus disease.

DETAILED DESCRIPTION:
This phase I study is designed to select patients with refractory and intractable disease. SLE patients with impaired visceral organ function and chronic exposure to glucocorticoid therapy are complicated by significant morbidity, frequent hospitalizations and high-risk of mortality. For participants in whom the indication is nephritis, active disease must be present despite at least 6 cycles of monthly pulse cyclophosphamide. Participants with extra-renal lupus need to fail 3 months of monthly cyclophosphamide. Patients who have an HLA matched sibling, will be offered allogeneic HSCT. Because of high transplant related toxicity and mortality in conventional myeloablative regimens, we will utilize a mini-conditioning regimen. To minimize GvHD, candidates must be 50 years old or younger and in vivo CAMPATH will be used in the conditioning regimen to deplete infused donor lymphocytes.

Peripheral Blood Stem Cell (PBSC) Harvest from Donor PBSC will be mobilized with G-CSF 10 mcg/kg/day (dose may be adjusted to 5-16 mcg/kg/day by PI for toxicity, e.g. flu-like symptoms) with stem cell collection beginning on day 4. Leukapheresis may be repeated up to three consecutive days.

1) If these criteria are not meet the patient (recipient) may not be treated.

1. CD34+ cell count >2.0 x106 CD34+ cells/kg recipient weight
2. Gram stein negative
3. Culture negative ( after 14 days)
4. Cell viability at time of final formulation in cyroprotectant media≥ 70% Conditioning Regimen Cyclophosphamide 50mg/kg/day x 4 days will be given IV over 1 hour in 500 cc of normal saline. If actual weight is < ideal weight, cyclophosphamide will be given based on actual weight. If actual weight is > ideal weight, cyclophosphamide will given as adjusted weight. Adjusted weight = ideal weight + 25% (actual weight minus ideal weight).

Mesna 50mg/kg/day will be given IV over 24 hours in 250 cc of normal saline or D5W starting 2 hours before the first cyclophosphamide dose. Weight base is calculated same as cyclophosphamide as above.

Hydration approximately 50-200cc/hour in adults should begin 6 hours before cyclophosphamide and continue until 24 hours after the last cyclophosphamide dose. Hydration rates need to be individually adjusted by daily weights to maintain dry weight count. BID weights will be obtained. Warning: Participants with renal insufficiency are prone to volume overload. Early institution of ultra filtration or dialysis is recommended. Three-way bladder irrigation may be needed for those participants who cannot tolerate fluid hydration during cyclophosphamide administration and for 24 hours after the last dose of cyclophosphamide. In patients on hemodialysis, cyclophosphamide will be given in the evening and hemodialysis will be performed in the morning daily until the last dose of cyclophosphamide is administered. Close coordination with nephrology service is required.

CAMPATH-1H 30mg/day x 2 days (no dose adjustment) will be given IV over 2 hours in 100 cc of normal saline. Premedication with acetaminophen 650mg and benadryl 50mg PO/IV will be given 30-60min before infusion. These medications can be repeated as needed. Solumedrol 1 gram will be given IV 30 min prior to CAMPATH-1H.

G-CSF 5 mcg/kg/day will be started on day 6 if engraftment has not occurred. It will be continued until absolute neutrophil count reaches at least 500/ul. The dose may be rounded up or down in order to not waste medication in the vial. NOTE: GCSF may be started earlier, e.g. day 0, per investigator's discretion.

Cyclosporine* will be started on day -3 at 200 mg po BID and adjusted by HPLC levels to between 150 - 250 or by toxicity (e.g., tremor, renal insufficiency, TTP, etc.). CSA will be continued for 2 months unless stopped for toxicity. If patient cannot tolerate oral cycloporine, intravenous cyclosporine continuous infusion (3mg/kg/24hours) and adjusted by levels can be used.

Mycophenolate mofetil (MMF)* 1g PO/IV q 12 hrs will be started on day -3 and continued for 6 months. The dosage will be adjusted and tapered off before stopping, unless toxicity mandates abrupt cessation. MMF will be adjusted by PI according to toxicity, GVHD, and donor engraftment or donor chimerism.

*Cyclosporine and MMF guidelines dosage and duration can be modified according to investigators discretion based on side effects, renal function, CBC and GVHD status.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Ages 18 to 50 years old.
* Meet at least 4 of 11 American College of Rheumatology (ACR) Classification criteria for SLE (see Appendix 1).
* Able to give informed consent.
* HLA matched sibling donor available.
* Meet one of following three:

  1. For lupus nephritis, participants must fail pulse cyclophosphamide (500 to 1000 mg/m2 monthly for a minimum of 6 months). Failure is defined as meeting criteria to be considered as BILAG (Appendix 4) renal category A. If indication for HSCT is nephritis, a renal biopsy must be obtained and document either class III or IV glomerulonephritis.
  2. For visceral organ involvement other than nephritis, participants must be BILAG cardiovascular/respiratory category A, vasculitis category A, or neurologic category A and must fail at least 3 months of oral or IV cyclophosphamide and be corticosteroid dependent. Steroid dependence being defined as at least 3 months of steroid therapy and inability to wean corticosteroid to less than 20 mg/day of prednisone or equivalent.
  3. For cytopenias that are immune mediated, participants must be BILAG hematologic category A. Participants must have an inability to maintain platelets > 15,000, an inability to prevent active bleeding without transfusion, an inability to maintain hemoglobin > 7.0, or an inability to prevent cardiovascular disease without transfusion. In addition, participants must fail corticosteroids (either oral prednisone > 0.5 mg/kg/day for more than 6 months or pulse methylprednisolone for at least one cycle of three days), be refractory to IVIG, and at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, mycophenolate mofetil 2 grams daily for more than 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months, danazol for at least 3 months, or splenectomy.

Recipient Exclusion Criteria:

* HIV positive.
* Ongoing malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the participant is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I or II breast cancer will be considered on an individual basis by the investigators doing the final screening for participant qualification.
* Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* DLCO < 45% of predicted unless attributed solely to active lupus.
* Resting LVEF < 40% unless due to active lupus.
* Known hypersensitivity to E. Coli derived proteins.
* Transaminases greater than 2 times normal unless due to active lupus.
* Any illness that in the opinion of the investigator would jeopardize the ability of the patient to tolerate this treatment.

Donor Inclusion Criteria

* Donor must be a HLA identical sibling or HLA matched cord blood donor.
* If donor is HLA matched sibling, donor must be > 18 years of age and less than 50years old.
* If multiple HLA matched donors are available, preference will be given to samesex, same CMV status, and nulliparous donor, or in the case of cord blood higher nucleated cell count.
* If donor is HLA matched cord blood, cord blood stem cells will be obtained from the New York Blood Center Cord Blood Registry (Tel 212-570-3230) which is an internationally recognized registry or, if a match is not available, from Stemcyte (626-821-9860) which is a commercial registry that specializes in minority donors or from National Marrow Donor Program (NMDP). One unit of HLA matched cord blood unit will be infused on day zero.

Donor Exclusion Criteria

* Physiologic age > 50 years old or <18 years old.
* HIV positive.
* Active ischemic heart disease or heart failure.
* Acute or chronic active hepatitis.
* Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the donor to tolerate stem cell collection.
* Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
* Positive pregnancy test.
* Positive ANA or anti-ds DNA.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* Major hematological abnormalities such as platelet count less than 150,000/ul, ANC less than 1000/ul.
* If donor is sibling must collect a minimum of 2. 106CD34+ cells/kg to proceed to Transplant.
* If donor is cord blood unit(s) then a minimum number of nucleated cells available must be more than 2 x 107 /kg. To achieve this number of nucleated cells, two units of HLA matched cord blood may be utilized. (Wagner JE Blood. 2005 Feb 1;105(3):1343-7)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Survival, disease free survival, number of relapses, organ function | Evaluation of response will be performed for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States